CLINICAL TRIAL: NCT01271374
Title: Changes in Central Aortic Pressure, Endothelial Function and Biomarkers in African Americans With Cardiometabolic Syndrome: Comparison of Amlodipine/Olmesartan Versus Hydrochlorothiazide/Losartan
Brief Title: Changes in Endothelial Function and Biomarkers in African Americans (AA) With Metabolic Syndrome
Acronym: AMORE
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: InVasc Therapeutics, Inc. (Industry)
Responsible Party: Bobby Khan, MD PhD, Atlanta Clinical Research Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AVR-2010-001
Record Dates: First submitted 2011-01-05; First posted 2011-01-06 (Estimated); Last update posted 2011-05-05 (Estimated); Status verified 2011-05

CONDITIONS: Hypertension
Keywords: African American; Hypertension; Cardiometabolic Syndrome
MeSH Terms: conditions — Hypertension; Metabolic Syndrome | interventions — Amlodipine Besylate, Olmesartan Medoxomil Drug Combination; Hydrochlorothiazide; Losartan; hydrochlorothiazide, losartan drug combination; Spironolactone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Hyzaar-Treatment Arm B (Active Comparator): Weeks 1-2: Hyzaar® 50/12.5 Weeks 3-14: Hyzaar® 100/25 Weeks 15-18: Azor® 10/40+HCTZ 25 Weeks 19-20: Azor® 10/40+HCTZ 25 + spironolactone 25 once daily
  Interventions: Drug: losartan and HCTZ
- Azor-Treatment A (Active Comparator): Weeks 1-2: Azor® 5/20 Weeks 3-14: Azor® 10/40 Weeks 15-18: Azor® 10/40+HCTZ 25 Weeks 19-20: Azor® 10/40+HCTZ 25 + spironolactone 25 once daily
  Interventions: Drug: amlodipine and olmesartan

INTERVENTIONS:
Drug: amlodipine and olmesartan — Weeks 1-2: Azor® 5/20 Weeks 3-14: Azor® 10/40 Weeks 15-18: Azor® 10/40+HCTZ 25 Weeks 19-20: Azor® 10/40+HCTZ 25 + spironolactone 25 once daily
  Other Names: Azor; Hydrochlorothiazide; Spironoloactone
  Arms: Azor-Treatment A
Drug: losartan and HCTZ — Weeks 1-2: Hyzaar® 50/12.5 Weeks 3-14: Hyzaar® 100/25 Weeks 15-18: Azor® 10/40+HCTZ 25 Weeks 19-20: Azor® 10/40+HCTZ 25 + spironolactone 25 once daily
  Other Names: Hyzaar; Azor; Hydrochlorothiazide; Spironolactone
  Arms: Hyzaar-Treatment Arm B

SUMMARY:
The purpose of the study is to compare the effects of Azor (a combination of amlodipine and olmesartan) with Hyzaar ( a combination of losartan and hydrochlorothiazide) on the thin lining on the inside of blood vessels. These cells help keep blood vessels healthy and blood pressure normal.

DETAILED DESCRIPTION:
Participants must be 18-75 years of age, African American, and have a combination of high blood pressure, insulin resistance (Type 2 Diabetes), low HDL cholesterol levels or obesity.

ELIGIBILITY:
Inclusion Criteria:

* African American
* Hypertension and one of the following:
* Fasting glucose > 100 mg/dl
* HgA1C> 6.0 %
* Plasma triglycerides >150
* HDL cholesterol < 40 mg/dl in men or < 50 mg/dl in women

Exclusion Criteria:

* History of Heart failure
* use of insulin
* non-dominant arm circ > 50 cm.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2010-04; Primary Completion 2011-06 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Change in Central Aortic Pressure (CAP) | 14 weeks
  The primary efficacy endpoints, defined as the change from baseline of Central Aortic Systolic Pressure (CAP) and the change in brachial artery reactivity (BART) via ultrasound testing, will be compared at the end of 14 weeks of randomized treatment.

SECONDARY OUTCOMES:
Blood pressure control | 25 weeks
  Secondary endpoints of percentage of subjects achieving BP goals will be analyzed using Cochran-Mentel-Haenzsel test.

CONTACTS AND LOCATIONS:
Overall Officials: Bobby V Khan, MD, PhD, Principal Investigator — Director, Atlanta Clinical Research Centers; Keith C Ferdinand, MD, Study Director — Atlanta Clinical Research Centers
Locations (1):
- Atlanta Clinical Research Center, Tucker, Georgia, United States